CLINICAL TRIAL: NCT07253597
Title: Effect of a Tactical Critical Thinking Intervention on Technical-tactical Decision-making in University Volleyball: A Quasi-experimental Study
Brief Title: Critical Thinking Volleyball Tactics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Édison Andrés Pérez Bedoya, PhD, Federal University of Vicosa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Volley_USB_TdeA
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Decision Making; Athletic Performance; Volleyball
Keywords: Tactical Critical Thinking Program; Volleyball; Team sports; Decision making; Technical-tactical skills

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, non-randomized, parallel assignment with two arms. Participants belong to one university men's volleyball programme and remain in a single arm for the entire study. One arm receives usual volleyball training enriched with the Tactical Critical Thinking Program (structured reflective pauses and guided questioning within game-based practice). The comparison arm continues with usual training only, without the structured reflective component. Both arms follow similar schedules, volumes and intensities of training. Outcomes are assessed at baseline and at the end of the intervention period to compare pre-post changes between arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPCT (Experimental): Participants in this arm attend their usual university volleyball practices enriched with the Tactical Critical Thinking Program. Training follows the regular team schedule (approximately three 90-minute sessions per week for 4 weeks) and is fully integrated into routine practice. The intervention adds game-based drills and small-sided games focused on serve, reception and spike, combined with brief, structured pauses. During these pauses, the coach guides players to analyse recent sequences, identify tactical problems, propose and justify alternatives and agree collective adjustments. A final phase of more open play emphasises applying these decisions, with prompts that foster metacognition. Training volume and physical workload are comparable to the comparison arm; the distinctive element is the structured critical-thinking and reflective-dialogue component.
  Interventions: Other: Tactical Critical Thinking Program plus usual volleyball training
- C-TPCT (Active Comparator): Participants in this arm attend their usual university volleyball practices without any added reflective component. Training follows the regular team schedule (approximately three 90-minute sessions per week for 4 weeks) and includes standard warm-up, physical preparation, technical drills and team play focused on serve, reception, spike and defensive actions, as determined by the coaching staff. Coaches do not implement the protocolised reflective pauses or guided questioning used in the experimental arm. Training volume, frequency and overall intensity remain comparable to those of the intervention arm, so that the main planned difference between groups is the absence of the structured critical-thinking and collaborative-reflection activities in this control condition.
  Interventions: Other: Usual volleyball training

INTERVENTIONS:
Other: Tactical Critical Thinking Program plus usual volleyball training — Behavioral intervention integrated into regular university men's volleyball practice. The program adds structured reflective pauses and guided questioning to usual training content (serve, reception, spike and team play). Sessions use game-based drills and small-sided games under modified constraints to elicit tactically demanding situations. After short sequences of play, the coach leads brief discussions in which players identify tactical problems, generate and justify alternatives and agree collective adjustments. A final phase of open play emphasises applying these decisions while promoting metacognitive reflection. Training frequency, duration and physical workload remain comparable to the control arm; the distinctive element is the protocolised critical-thinking and collaborative-reflection component.
  Arms: TPCT
Other: Usual volleyball training — Behavioral condition consisting of the team's standard university men's volleyball training program with no added reflective component. Sessions include warm-up, general physical preparation, technical drills for serve, reception, spike and defence, positional work and team play under normal coaching practice. Coaches do not apply the structured reflective pauses or guided questioning protocol used in the experimental arm. Training schedule, session duration and general intensity are maintained as similar as possible to the intervention arm so that the principal difference between arms is the absence of the Tactical Critical Thinking Program.
  Arms: C-TPCT

SUMMARY:
This quasi-experimental study will examine whether a Tactical Critical Thinking Program (TPCT) can improve technical-tactical decision-making in university volleyball players compared with usual training. In many university teams, practice is dominated by repetitive technical drills and coach-centred instruction, with limited opportunities for players to analyse the game, discuss options with teammates, or reflect critically on their decisions.

The study compares two groups of adult male volleyball players from a university-level programme in Colombia. The intervention group completed a 4-week Tactical Critical Thinking Program integrated into regular volleyball practice, while the comparison group continued with their usual training routines, without structured reflection or guided questioning. The TPCT uses representative game-based tasks, short planned pauses for group discussion, and questions that prompt players to identify tactical problems, generate alternative solutions, justify their choices, and adjust strategies collectively.

All participants assessed before and after the 4-week period. Assessments included validated technical skill tests for serve, reception and spike, and standardised small-sided games (4 vs 4) recorded on video. Trained observers coded each action to calculate decision-making indices for the three key skills, expressing the proportion of tactically appropriate decisions during play.

The primary aim was to determine whether adding structured tactical reflection and critical thinking activities to volleyball practice produces greater improvements in decision-making than usual training alone. A secondary aim was to explore whether the TPCT also enhances technical execution. Findings are expected to inform coaches and physical education professionals about how to design cognitively enriched, game-representative training for university team sports.

DETAILED DESCRIPTION:
This interventional study evaluates the effect of a Tactical Critical Thinking Program (PTPC, by its Spanish acronym) on technical-tactical decision-making in university volleyball. The study uses a quasi-experimental, non-randomized, parallel-group design with intentional allocation. One group receives regular volleyball training enriched with the PTPC, and a comparison group continues with usual practice routines without structured reflective spaces.

The setting is a university men's volleyball programme in Cartagena, Colombia. Eligible participants are adult male players who belong to the university team, have regular training experience, are medically cleared for full participation and can attend the planned training and assessment sessions. Exclusion criteria include any current injury or medical restriction for sport participation and an inability to comply with the intervention schedule.

The PTPC integrates critical thinking and collaborative reflection into representative volleyball practice. Across approximately 12 sessions, embedded within normal team training, each session follows a stable pedagogical sequence. An initial brief activation phase clarifies the tactical focus of the day (for example, organisation of reception, serve-receive-attack connections or spike decision-making) and invites players to identify recurrent problems and shared objectives. The central phase consists of game-based drills and small-sided games that manipulate numerical relations, court spaces and rules to expose players to tactically demanding situations involving serve, reception, spike and defensive actions. Within this central phase, the coach introduces short, preplanned pauses in which players analyse recent sequences and discuss what is working, what is limiting performance, which technical resources they use or lack, and which tactical or positional adjustments they propose. A final phase of more open play under full rules emphasises the application and refinement of the agreed tactical adjustments and promotes metacognitive reflection on why certain options are chosen and how they relate to collective strategy.

The comparison group follows the usual training programme designed by the coaching staff. This programme includes warm-up, physical preparation, technical drills and team game play, but it does not include the protocolised reflective pauses or the guided questioning structure that characterises the PTPC. Training volume, frequency and general intensity remain as comparable as possible between groups so that the main planned difference is the presence or absence of the structured critical-thinking component.

Outcomes focus on technical-tactical performance in serve, reception and spike. Technical execution is assessed through a standardised battery of volleyball skill tests that quantify accuracy and consistency for each action using target zones and scoring criteria based on established methodological references. Tactical decision-making is assessed during standardised small-sided games (for example, 4 vs 4) on a regulation court under official rules. Games are video recorded, and trained observers code each serve, reception and spike as tactically appropriate or inappropriate according to predefined criteria (such as serving to vulnerable zones, directing reception to an optimal setting area, or attacking into uncovered spaces). For each player and each skill, a decision-making index represents the proportion of appropriate actions out of the total number of observed actions.

Assessments take place in the week immediately before the intervention period and in the week after its completion. Data collection also includes basic sociodemographic and anthropometric information (for example, age, training experience, body mass, height and body mass index) in order to characterise the sample and, if necessary, use these variables as covariates. Observers receive training in systematic notation of volleyball actions, and inter-observer agreement is checked prior to formal coding to ensure acceptable reliability.

Data management relies on anonymised participant codes and secure storage of datasets and video material. Statistical analysis describes the sample with means, standard deviations, medians and interquartile ranges as appropriate. Pre-post changes in decision-making indices and technical scores are analysed within each group, and differences in change between the PTPC and comparison groups are examined with standard parametric or non-parametric tests according to distribution, complemented by effect sizes and 95% confidence intervals. The level of significance is set at 0.05, and interpretation acknowledges the quasi-experimental, non-randomized nature of the design.

The study aims to provide evidence on whether embedding a structured critical-thinking programme into routine volleyball practice optimises decision-making and technical performance, and whether this model offers a transferable framework for other team sports and educational contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* University volleyball player enrolled in the participating programme in Medellín, Colombia
* Regular participation in team training (at least two organised sessions per week before study enrolment)
* Medically cleared and physically able to take part in full volleyball training and match play
* Availability to attend the majority of scheduled intervention and assessment sessions over the ≈ 4-week study period
* Provision of written informed consent

Exclusion Criteria:

* Current musculoskeletal injury or medical condition that limits safe participation in volleyball training or matches
* Any medical contraindication to high-intensity intermittent exercise as reported by the participant or team medical staff
* Planned absence that would prevent attendance at baseline or post-intervention assessments or more than 20% of training sessions
* Concurrent participation in another structured intervention specifically targeting tactical decision-making or psychological skills in volleyball
* Withdrawal of consent at any point before completion of post-intervention assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change in decision-making index during standardized game situations | Baseline (week 0) and immediately post-intervention (within 1 week after the last training session; total intervention period ≈ 4 weeks)
  Decision-making index during standardized small-sided volleyball games (for serve, reception and spike). The index represents the proportion of tactically appropriate actions out of the total number of coded actions in 4 vs 4 games on a regulation court. Actions are coded from video by trained observers using predefined criteria (for example, serve to vulnerable zones, reception directed to an optimal setting area, spike to uncovered spaces). Higher scores indicate a greater proportion of tactically appropriate decisions. Analyses compare change from baseline to post-intervention between the Tactical Critical Thinking Program arm and the usual-training control arm.

SECONDARY OUTCOMES:
Change in decision-making index for serve | Baseline (week 0) and immediately post-intervention (within 1 week after the last training session; total intervention period ≈ 4 weeks)
  Decision-making index for serve during standardized 4 vs 4 games. Each serve is coded as tactically appropriate or inappropriate according to predefined criteria (for example, direction and depth toward vulnerable reception zones). The index is the proportion of appropriate serves out of all serves performed by each player. Higher values indicate better serve-related tactical decision-making. Change from baseline to post-intervention is compared between arms.
Change in decision-making index for reception | Baseline (week 0) and immediately post-intervention (within 1 week after the last training session; total intervention period ≈ 4 weeks)
  Decision-making index for reception during standardized 4 vs 4 games. Each reception is coded as tactically appropriate or inappropriate according to predefined criteria (for example, directing the ball to an optimal setting zone or player). The index is the proportion of appropriate receptions out of all receptions performed by each player. Higher values indicate better reception-related tactical decision-making. Change from baseline to post-intervention is compared between arms.
Change in decision-making index for spike | Baseline (week 0) and immediately post-intervention (within 1 week after the last training session; total intervention period ≈ 4 weeks)
  Decision-making index for spike during standardized 4 vs 4 games. Each spike is coded as tactically appropriate or inappropriate based on predefined criteria (for example, attacking into uncovered spaces or exploiting blocking mismatches). The index is the proportion of appropriate spikes out of all spikes performed by each player. Higher values indicate better spike-related tactical decision-making. Change from baseline to post-intervention is compared between arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de San Buenaventura - Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results (decision-making indices, technical skill test scores and basic demographic variables such as age and playing experience) are available to other researchers for academic, non-commercial use. No video files or direct identifiers are shared. Data access depends on a reasonable research proposal and the signing of a data use agreement that prohibits re-identification or data linkage with other identifiable sources.
Supporting Information: Study Protocol, SAP
Time Frame: IPD are available starting approximately 6 months after publication of the main results paper and remain available for at least 5 years thereafter, or as long as the dataset is curated by the investigators.
Access Criteria: Researchers send a brief proposal describing objectives, methods and requested variables to the corresponding author. Proposals are reviewed by the study team and, when applicable, by the institutional ethics committee. Once approved, data are shared in de-identified format under a data use agreement that limits use to the approved project, forbids attempts at re-identification and excludes commercial use.